CLINICAL TRIAL: NCT04470089
Title: A Multi-center, Randomized, Placebo-controlled, Double-blind, Dose-finding Clinical Trial Investigating the Short-term Relief of Symptoms of Acute Pharyngitis Such as Throat Soreness Pain and Difficulty to Swallow by Treatment With Three Different Doses of MYRAMISTIN™ Oromucosal Spray
Brief Title: A Clinical Trial Investigating the Short-term Relief of Symptoms of Acute Pharyngitis by Treatment With Three Different Doses of MYRAMISTIN™ Oromucosal Spray
Acronym: MIRA1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to the COVID situation by end of 2021 and therfore limited recruitment of patients diagnosis "acute pharyngitis" the study was terminated.
Sponsor: Megainpharm GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MIRA1
Record Dates: First submitted 2020-05-19; First posted 2020-07-14 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Acute Pharyngitis
MeSH Terms: interventions — miramistin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Myramistin 0.005% (Experimental)
  Interventions: Drug: Myramistin
- Myramistin 0.01% (Experimental)
  Interventions: Drug: Myramistin
- Myramistin 0.02% (Experimental)
  Interventions: Drug: Myramistin
- Placebo (Placebo Comparator)
  Interventions: Drug: Myramistin

INTERVENTIONS:
Drug: Myramistin — Oromucosal application

SUMMARY:
In this multi-center, randomized, placebo-controlled, double-blind stuy in which patients with acute pharyngitis will receive Myramistin™ / Placebo, which is provided as a spray. Patients will be randomised at Visit 1 on a 1:1:1:1 basis to one of the three MyramistinTM doses (0.005%, 0.01% and 0.02%) or placebo. The trial duration for an individual patient is 72 hours.

The primary objective is to evaluate the short-term efficacy of different MyramistinTM doses (0.005%, 0.01% and 0.02%) compared to placebo in the symptomatic treatment of acute pharyngitis.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female at the ages of 18 to 75 years
2. Body Mass Index (BMI): 18-31 kg/m2
3. Willing and able to give informed consent
4. Clinically diagnosed acute pharyngitis.
5. Onset of symptoms of acute pharyngitis within the past 48 hours prior to Visit 1
6. Symptoms of acute pharyngitis such as sore throat and difficulty to swallow
7. Sore throat pain intensity scored as at least 60 mm on a 0-100 mm VAS (Visual Analogue Scale) Sore Throat Pain Intensity Scale (STPIS)
8. Difficulty in swallowing of at least 60 mm on a 0-100 mm VAS Difficulty Swallowing Scale (DSS)
9. Tonsillo-Pharyngitis Assessment (TPA) ≥ 6 on 21-point TPA- scale
10. Absence of Group A Streptococcus as confirmed by a rapid swab test before randomization
11. McIsaac - Score <3
12. Willing to stay in the trial center for at least 2 hours (maximum 3 hrs) after the first dose and return after 72 hours treatment on Day 4
13. Willing not to take anything by mouth excluding the investigational medical product (IMP) and / or unable to abstain from smoking during the stay in the trial center. Drinking of water is allowed.
14. Female patients must have

    * either a negative pregnancy test at Visit 1 and practicing a reliable method of contraception used consistently and correctly (including oral contraceptives, hormone implant, intrauterine device), or
    * must be postmenopausal (not spontaneous menstrual periods for at least 6 months) or
    * must be surgically sterile (tubal ligation or removal of ovaries or uterus)

Exclusion Criteria:

1. Patients with strong suspicion of Group A streptococcus infection. Either swab test is positive OR McIsaac Score ≥ 3 points
2. Presence of signs or symptoms of any acute infection for which treatment with antibiotics is mandatory and/or should not be postponed; i.e. accompanied fever (> 38°C at Visit 1) and/or - if visually identified pharyngeal - presence of seropurulent, purulent, fibro serous or fibrinous exudate from the pharyngeal mucosa
3. Patients with allergies or bronchial asthma who have a history of exacerbations within 30 days prior to trial inclusion
4. The use of any systemic analgesics / local analgesics in the throat area (e.g. Acetyl Salicylic Acid = ASA > 100 mg) during the trial or within 12 hours prior first study medication application. Exception Paracetamol: intake of Paracetamol is allowed up to 6 hours before first application of IMP
5. The use of systemic antibiotics / local antibiotics in the throat area during the trial and within the previous 7 days prior to Visit 1
6. The use of any systemic or local (i.e. in the throat area) antihistamines started within 2 weeks prior to Visit 1
7. The use of any systemic anti-inflammatory drug / local anti-inflammatory drug in the throat area (e.g. non-steroidal anti- inflammatory drugs or glucocorticoids) during the trial or within 12 hours prior to first IMP application
8. The use of local anaesthetics for treatment of sore throat during the trial or within 12 hours prior to first IMP application
9. The use of any other 'sore throat medication' (e.g. lozenges, drops, sprays, decongestants) or other 'cold medication' that could interfere the trial results within the previous 12 hours prior to first study medication application
10. Major wounds of the mouth and throat
11. Immunodeficiency disorders (e.g. organ transplantation, HIV infection)
12. Existing cardiac, haematological, hepatic, renal, gastrointestinal, metabolic and / or pathological findings, which might interfere with the drug's safety, tolerability and / or absorption according to the judgement of the Investigator
13. Any neurological or psychiatric conditions, which might give the impression that the patients will not comply with the protocol and trial needs
14. Patients with history (previous 5 years) or present condition of any malignancy
15. Known hypersensitivity to any ingredient of MyramistinTM
16. Previous participation in the trial
17. Parallel participation in any other trial during the previous 90 days before screening
18. History of alcohol or drug abuse
19. Known or suspected of being unable to comply with the clinical trial protocol (e.g. no permanent address, history of drug abuse, known to be non-compliant or presenting an unstable psychiatric history)
20. Legal incapacity and / or other circumstances rendering the patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Pain Intensity Differences | 2 hours
  The primary endpoint is the Summed Pain Intensity Differences (SPID-2Pain), defined as Pain Intensity Differences (PID) summarized over the time course of 2 hours after first application on Day 1 (Baseline). The sum is calculated over the time-weighted differences from each measured time point to baseline after dosing using the 100mm Visual Analogue Scale (VAS) Sore Throat Pain Intensity Scale (STPIS).

SECONDARY OUTCOMES:
Pain Intensity Differences | 72+/-2 hours
  Pain Intensity Differences (PID) is summarized at different defined timepoints after first application on Day 1 (Baseline). The sum is calculated over the time-weighted differences from each measured time point to baseline after dosing using the 100mm VAS Sore Throat Pain Intensity Scale (STPIS).
Difficulty to Swallow Differences | 72+/-2 hours
  SPID2-Swallow calculated analogously to the primary endpoint (including sensitivity analysis) using the Difficulty Swallowing Scale (DSS), furthermore it is calculated on different predefined timepoints.
Time to Pain Relief | 72+/-2 hours
  Time to 30% and 50% pain relief (30% and 50% reduction in STPIS) compared to baseline.
Time to relief in Difficulty to Swallow | 72+/-2 hours
  Time to 30% and 50% relief in difficulty in swallowing (30% and 50% reduction in DSS) compared to baseline.
Percentage of symptom free patients | 72+/-2 hours
  * in throat pain at Visit 2 (STPIS=0)
  * in difficulty in swallowing at Visit 2 (DSS=0)
  * in throat pain and difficulty in swallowing at Visit 2 (STPIS=0 and DSS=0 - defined as complete
Tonsillo-Pharyngitis Assessment Scale | 72+/-2 hours
  Change in Tonsillo-Pharyngitis Assessment (TPA) sum-score and single symptom scores from baseline to Visit 2 Variables (findings like e.g. oral temperature, oropharyngeal colour, size of tonsilles etc.) presented are rated using the values 0, 1, 2 or 3 (points). The points are added together to make a TPA that can range from 0 to 21 points. Pharyngitis is present if a total score of ≥6 is obtained.

OTHER OUTCOMES:
Safety Endpoints | 72+/-2 hours
  Type, frequency, severity and assessment of drug relationship of reported adverse events and will be descriptively evaluated and compared between treatment arms.
Tolerability Endpoints | 72+/-2 hours
  Treatment differences in global assessment of tolerability will be tested using the Wilcoxon test adjusted for center (Van Elteren test) separately for patient and Investigator assessment.

CONTACTS AND LOCATIONS:
Locations (12):
- Austria (3):
  - KAR, Vienna
  - MUW, Vienna
  - Zentrum für Klinische Studien, Vienna
- Germany (9):
  - Practive, Berlin
  - Practice, Cologne
  - Practice, Duisburg
  - Practice, Fulda
  - Practice, Goch
  - Practice, München
  - Practice, Neuenhagen
  - Practice, Rosenheim
  - Practice, Wuppertal